CLINICAL TRIAL: NCT04665284
Title: Safety And Efficacy Of Empagliflozin In Pakistani Muslim Population With Type Ii Diabetes Mellitus
Acronym: SAFE-PAK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Getz Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GTZ-DM-001-19
Record Dates: First submitted 2020-11-27; First posted 2020-12-11 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Type II Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin (Experimental)
  Interventions: Drug: Empagliflozin
- Usual Care Group (Active Comparator)
  Interventions: Drug: Usual care group

INTERVENTIONS:
Drug: Empagliflozin — Group A: Empagliflozin 10/25 mg once daily with or without antidiabetic drugs
  Other Names: Group A
  Arms: Empagliflozin
Drug: Usual care group — Group B: usual care group but without Empagliflozin with adjustment of therapy as the standard of care
  Other Names: Group B
  Arms: Usual Care Group

SUMMARY:
To compare the safety and efficacy of empagliflozin versus other treatments in Pakistani Muslim population with type II diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes is the one of the most common non-communicable diseases affecting 425 million adults worldwide. This figure is expected to rise to 629 million by the year 2045.1 90% of the diabetic population has type 2 diabetes. 2 As of 2018, more than 500 million individuals are residing with type 2 diabetes mellitus globally. 3 In Pakistan, the situation is similarly alarming. According to a recent survey, 16.98% of the Pakistani population has diabetes.4 The primary target of therapy in diabetes mellitus is optimum blood glucose control. In case of type 2 diabetes, this is achieved by a combination of oral hypoglycemic agents and injectable drugs with insulin as a last resort.

A number of oral agents targeting various sites of action are available. Sodium-glucose cotransporter-2 (SGLT2) inhibitors are newer class of drugs that have been introduced. They have a unique mechanism of action. By acting at the sodium glucose co-transporter, they block the reabsorption of glucose leading to an increase in urinary glucose excretion and lowering of plasma glucose.5 This action is completely independent of the beta cell function. There are several theoretical advantages to this approach. In addition to lowering blood glucose, the urinary glucose excretion results in loss of calories and weight reduction and the associated osmotic diuretic effect can aid in lowering blood pressures.6,7 Numerous studies have demonstrated a favorable risk benefit ratio of empagliflozin as monotherapy8 as well as add-on therapy to other hypoglycemic agents.9,10,11,12 They also have additional cardiovascular benefits with several studies documenting a reduction in mortality.13,14 Moreover, the sodium glucose co-transporters also demonstrated a reduction in the onset and worsening of nephropathy and preservation of renal function.15 This effect is not restricted to empagliflozin alone, as other drugs in the class have also demonstrated this benefit.16 Empagliflozin with its novel mechanism of action has its own set of side effects. Increased urinary glucose losses lead to a higher proportion of urinary tract infections and genital tract infections. This has been evidenced in various studies.17 The osmotic diuresis that benefits in lowering blood pressures at one end, also predisposes the patients to volume depletion.Empagliflozin, one of the three drugs from this class, approved by the FDA for treatment of type 2 diabetes. According to the recent ADA and the EASD guidelines, they have become an essential component of the algorithm recommended for managing type 2 diabetes.18 The recently published consensus statement by the South Asian Federation of Endocrine Societies has incorporated sodium glucose co-transporter 2 inhibitors in the treatment of patients with type 2 diabetes as monotherapy in patients who are intolerant to or have any contraindication to metformin therapy. Additionally, drugs belonging to this class are also recommended as combination therapy with other oral hypoglycemic agents as well as insulin.19 Empagliflozin, however, has not been studied in the Pakistani population as yet. The main aim of this study is to establish the efficacy and safety of empagliflozin in optimum control of blood sugar in type 2 diabetes. This is the first study of its kind being performed in the Pakistani population.

ELIGIBILITY:
Inclusion Criteria:

* Pakistani muslim male / female, type 2 diabetic patient having age from 18 years to 75 years
* Patient who give informed consent voluntarily
* BMI ≤45 kg/m2
* Glycosylated hemoglobin of 7 - ≤10%

Exclusion Criteria:

* Patients who are on empagliflozin treatment
* Indication of liver disease, defined by serum levels of either alanine aminotransferase, aspartate aminotransferase, and alkaline phosphatase above 3 times upper limit to normal
* Estimated glomerular filtration rate (eGFR) <45 mL /min /1.73m2
* History of recurrent urinary tract infection (UTI) and/or past 3 months' history of UTI and its treatment
* Patients with positive urine culture for UTI at the time of screening
* Patients who have been admitted to the hospital in the past 3 months for diabetic ketoacidosis (DKA) and hyperosmolar hyperglycemic state
* Patients with past 3 months' history of fungal infection and its treatment
* History of blood dyscrasias or any disorders causing haemolysis or unstable red blood cell
* History of benign prostate hyperplasia
* Any acute coronary syndrome, stroke and/or transient ischemic attack (TIA) in the previous 3 months
* Any contraindication for patients to Biguanides, Sulfonylureas, DPP-IV inhibitors, SGLT-2 Inhibitors
* Treatment with anti-obesity drugs or any other treatment leading to unstable body weight
* Patients with past 6 weeks treatment history with systemic steroids or thyroid hormones or any other uncontrolled endocrine disorder except T2DM
* Pre-menopausal women who are nursing or pregnant or are of childbearing potential and not practicing an acceptable method of birth control
* Any other clinical condition that would jeopardize patients safety while participating in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-28 (Actual)

PRIMARY OUTCOMES:
Number of participants reported adverse events | 24 weeks
  Number of participants reported adverse events such as Hypoglycemic events, Hypotension, Dehydration, Urinary tract infection, Diabetic Ketoacidosis, Fungal infection or any other

SECONDARY OUTCOMES:
Frequency of participants achieved HbA1c level <7% | 24 weeks
  Frequency of participants achieved HbA1c level <7%
Frequency of participants achieved FBS level within normal range | 24 weeks
  Frequency of participants achieved FBS level within normal range

OTHER OUTCOMES:
Number of participants reduces weight during the therapy | 24 weeks
  Number of participants reduces weight during the therapy or mean reduction in weight overtime
Number of participants reduces BMI level as per WHO Asian classification during the therapy | 24 weeks
  Number of participants reduces BMI or mean reduction in BMI overtime
Number of participants reduces Waist circumference during the therapy | 24 weeks
  Number of participants reduces Waist circumference or mean reduction in BMI overtime
Number of participants changes systolic blood pressure and diastolic blood pressure during the therapy | 24 weeks
  Number of participants reduces systolic blood pressure and diastolic blood pressure or mean reduction in systolic blood pressure and diastolic blood pressure overtime
Number of participants changes LDL level and HDL Level during the therapy | 24 weeks
  Number of participants reduces LDL level and HDL Level or mean reduction in LDL level and HDL Level overtime
Mean score of diabetes mellitus quality of life | 24 weeks
  The instrument provides an overall scale score, as well as two subscale scores for 1) satisfaction with treatment, 2) adherence with Self Care Regimen. 15 Items are scored on a 5-point Likert scale and are of two general formats.One format asks about the frequency of negative impact of diabetes itself or of the diabetes treatment and provides response options from 1 (never) to 5 (all the time). The second format asks about satisfaction with treatment and quality of life and is scored from 1 (very satisfied) to 5 (very dissatisfied). Higher scores on DQOL items and subscales are, therefore, negatively valenced, indicating problem frequency or dissatisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: A H Aamir, Principal Investigator — Post Graduate Medical Institute
Locations (11):
- Pakistan (11):
  - Balochistan Medical Center, Quetta, Balochistan
  - Lady Reading Hospital, Peshawar, Khyber Pakhtunkhwa
  - Post Graduate Medical Institute, Peshawar, Khyber Pakhtunkhwa
  - Hanif Medical Center, Islamabad, Punjab Province
  - Shifa International Hospital, Islamabad, Punjab Province
  - Diabetes Institute of Pakistan, Lahore, Punjab Province
  - Jinnah Hospital, Lahore, Punjab Province
  - National Defence Center, Lahore, Punjab Province
  - Al-Khaliq Hospital, Multan Khurd, Punjab Province
  - Fatimiyah Hospital, Karachi, Sindh
  - National Institute of Cardiovascular Disease, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aamir AH, Raja UY, Qureshi FM, Asghar A, Mahar SA, Ahmed I, Ghaffar T, Zafar J, Hasan MI, Riaz A, Raza SA, Khosa IA, Khan J, Baqar JB. Safety and efficacy of Empagliflozin in Pakistani Muslim patients with type 2 diabetes (SAFE-PAK); a randomized clinical trial. BMC Endocr Disord. 2022 Nov 28;22(1):295. doi: 10.1186/s12902-022-01213-1. PMID 36443769